CLINICAL TRIAL: NCT04202250
Title: Comparison of the Efficacy of Single-port Open-ended Catheter and Closed-end Multiport Catheters for Continuous Femoral Nerve Blockade for Postoperative Analgesia in Patients Undergoing Knee Arthroplasty
Brief Title: The Efficacy of Continuous Femoral Nerve Catheter Orifice Configuration for Postoperative Analgesia in Knee Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gulhane School of Medicine (Other)
Responsible Party: Principal Investigator, Mehmet Burak Eşkin, Assistant Professor, Gulhane School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 19/397
Record Dates: First submitted 2019-12-16; First posted 2019-12-17 (Actual); Last update posted 2020-05-18 (Actual); Status verified 2020-05

CONDITIONS: Anesthesia; Catheter Blockage; Knee Arthropathy; Pain, Postoperative
Keywords: femoral nerve catheter; Total Knee Arthroplasty; Catheter tips configurations; continuous nerve block
MeSH Terms: conditions — Pain, Postoperative | interventions — Population Groups

STUDY DESIGN:
Intervention Model Description: The patients will be randomized to the catheter tip configuration as CEMP (closed-ended multiport catheter) group and OESP (open-ended single port catheter) group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CEMP (closed-ended multiport catheter) group (Active Comparator): closed-ended multiport femoral nerve catheter will be included in the patients undergoing total knee arthroplasty surgery for postoperative analgesia
  Interventions: Procedure: CEMP (closed-ended multiport catheter) group
- OESP (open-ended single port catheter) group (Active Comparator): open-ended single port femoral nerve catheter will be included in the patients undergoing total knee arthroplasty surgery for postoperative analgesia
  Interventions: Procedure: OESP (open-ended single port catheter) group

INTERVENTIONS:
Procedure: CEMP (closed-ended multiport catheter) group — After sterile preparation and large inguinal crease draping, with the US probe in a sterile sleeve or cover , we will proceed to hydrolocalization with 5-10 mL 5% dextrose in order to open the space between the femoral nerve and the superior part of the ilio-psoas muscle. The Contiplex® FX Non-Stimulating Tuohy Set, 17Ga. x 3½ inches. the Non-Stimulating Needle and the closed-tip multiport catheter will be then inserted under control and its position assessed between the femoral nerve and the superior aspect of the ilio-psoas muscle. Some aliquots of 5% dextrose will inject to confirm correct dispersal of the solution along the femoral nerve. The catheter will be tunnelled subcutaneously.A patient-controlled analgesic device will be attached to the catheter for postoperative analgesia. continuous peripheral nerve patient-controlled analgesia is as follows: 0.125% bupivacaine; hourly infusion: 4 ml / hour, pca dose (bolus): 5 ml / hour, lock-up time: 30 min, 4-hours limit: 30 ml.
  Arms: CEMP (closed-ended multiport catheter) group
Procedure: OESP (open-ended single port catheter) group — After sterile preparation and large inguinal crease draping, with the US probe in a sterile sleeve or cover , we will proceed to hydrolocalization with 5-10 mL 5% dextrose in order to open the space between the femoral nerve and the superior part of the ilio-psoas muscle. The Contiplex® FX Non-Stimulating Tuohy Set, 17Ga. x 3½ inches. the Non-Stimulating Needle and the open-ended catheter will be then inserted under control and its position assessed between the femoral nerve and the superior aspect of the ilio-psoas muscle. Some aliquots of 5% dextrose will inject to confirm correct dispersal of the solution along the femoral nerve. The catheter will be tunnelled subcutaneously. A patient-controlled analgesic device will be attached to the catheter for postoperative analgesia. continuous peripheral nerve patient-controlled analgesia is as follows: 0.125% bupivacaine; hourly infusion: 4 ml / hour, pca dose (bolus): 5 ml / hour, lock-up time: 30 min, 4-hours limit: 30 ml.
  Arms: OESP (open-ended single port catheter) group

SUMMARY:
Femoral nerve catheter for postoperative analgesia will be included in the adult patients undergoing total knee arthroplasty included in the study. These patients will be randomized to the catheter tip configuration as CEMP (closed-ended multiport catheter) group and OESP (open-ended single port catheter) group. Patient controlled analgesia device will be attached to the peripheral nerve catheter of these patients. Demographic data of the patients , the number of pushing the button the amount of bolus dose given, and the total dose given in the patient controlled anesthesia device, the need for additional analgesia and the amount, pain scores, complications will be recorded for three days postoperatively. Records will be compared statistically.

DETAILED DESCRIPTION:
Ethics committee approval was received on 10 December 2019, numbered 19/397. The study was planned to include 90 adult patients undergoing total knee arthroplasty at Gülhane Training and Research Hospital between 10 December 2019 and April 2020. Continue femoral nerve catheter for postoperative analgesia will be included in the patients included in the study. These patients will be randomized to the catheter tip configuration as CEMP (closed-ended multiport catheter) group and OESP (open-ended single port catheter) group. Patient controlled analgesia device will be attached to the peripheral nerve catheter of these patients. Demographic data of the patients who have placed an femoral nerve catheter and used the catheter successfully for three days postoperatively, the number of pushing the button, the amount of bolus dose given and the total dose given in the patient controlled anesthesia device,the amounts of need for additional analgesia and pain scores(Numeric rating Scale), complications will be recorded for three days postoperatively. Records will be compared statistically.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) Score I-III
* upper extremity surgery

Exclusion Criteria:

* emergency surgery,
* secondary surgery,
* chronic pain treatment
* pregnancy,
* any contraindication to peripheral nerve blockade,
* pre-existing peripheral nerve neuropathy,
* allergy to LA (study medications),
* ASA score ≥ 4,
* neurologic or neuromuscular disease,
* psychiatric disease,
* renal failure,
* hepatic failure,
* NSAID contraindication,
* inability to use a patient controlled analgesia (PCA) device,
* infection at the injection site
* withdrawal of consent.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2019-12-10 (Actual); Primary Completion 2020-04-12 (Actual); Study Completion 2020-05-10 (Actual)

PRIMARY OUTCOMES:
numeric rating scale (NRS) | three days postoperatively
  Pain 0 (no pain) to 10 (worst pain imaginable), ranging from a numeric rating scale (NRS)
use of patient control analgesia | three days postoperatively
  The number of PCA button presses, the total amount of local anesthetics applied
complications related to opioids | three days postoperatively
  Nausea, Vomiting, Itching, Constipation, Difficulty in urination, Difficulty in Concentration,
the requirement for additional analgesia | three days postoperatively
  Additional analgesic dexketoprofen (trometamol) 50 mg / 2 ml will be administered intravenously as rescue analgesia to patients with an NRS score above 3 and recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Mehmet B EŞKİN, M.D., Study Director — Gulhane Training and Research Hospital; Ayşegül Ceylan, Principal Investigator — Gulhane Training and Research Hospital
Locations (1):
- Gulhane Training and Research Hospital, Ankara, Keçiören, Turkey (Türkiye)